CLINICAL TRIAL: NCT01770561
Title: Feasibility Study to Assess Performance of an Integrated Sensor and Infusion Set. TRIAL II
Brief Title: Feasibility Study of an Integrated Sensor and Infusion Set
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes R&D Denmark (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CER269
Record Dates: First submitted 2012-08-15; First posted 2013-01-18 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Integrated sensor and infusion set. (Experimental): All subjects must have been previously diagnosed Type 1 Diabetics and being used to sensor augumented pumps
  Interventions: Device: Integrated sensor and infusion set.

INTERVENTIONS:
Device: Integrated sensor and infusion set. — Change patients from current devices to the Integrated sensor and infusion set.

SUMMARY:
The purpose of this study is to collect performance data on the integrated sensor and infusion set during 3 days of use and demonstrate performance adequacy of the Integrated sensor and infusion set with glucose sensing and insulin delivery functionalities. The hypothesis of this study is that having the infusion of insulin in close proximity to the sensor does not interfere with the sensor accuracy.

DETAILED DESCRIPTION:
Sensor clinical accuracy will be evaluated based on the following parameters: Mean ARD (absolute relative difference), median ARD, Clarke Grid Analysis. Meter BG values will be used as reference. Descriptive statistics will be used to assess non-inferiority of the Integrated sensor and infusion sets sensors compare to control Enlite sensors.

Insulin delivery functionality will be evaluated based on BG profiles obtained during peri-prandial periods during which BG measurements will be performed at 15, 20, 30 min intervals according to a SMBG schedule. Post-prandial pharmacodynamic profiles will be analyzed to demonstrate the effect of insulin delivered using the Integrated sensor and infusion set. Specifically, rise in glucose levels followed by their fall will be used as an indication that insulin was delivered and absorbed. Post-prandial BG areas under the curve (AUC), Tmax (time to maximum rise of BG), and Cmax (maximum post-prandial BG) values will be calculated for each meal (breakfast, lunch, and dinner) consumed during both inpatient days and compared. Intra - and inter-subject mean values and standard deviations will be calculated. Paired and unpaired T-tests will be used to evaluate statistical significance.

Longevity of device performance will be assessed by comparing the listed parameters obtained during two inpatient days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 21-70 years of age at time of screening
2. Subject has a clinical diagnose of type 1 diabetes, as determined by investigator
3. Subject has one or more established insulin-to-carbohydrate ratios
4. Subject has one or more established insulin correction ratios
5. Subject is currently using a Medtronic insulin pump and has been so for a minimum of 3 months at time of enrollment.
6. Subject has been using insulin for more than one year.
7. Subject is willing to wear two pumps, one sensor, one infusion set and one Integrated sensor and infusion set at one time (first night).
8. Subject is willing to perform frequent SMBGs during Visits 3 and 4.
9. Subject is in good general health without other acute or chronic illnesses

Exclusion Criteria:

1. Subject is pregnant or lactating (if female), as self-declared by patient
2. Subject plans to become pregnant during the course of the study
3. Subject is unable to tolerate tape adhesive in the area of sensor placement
4. Subject has any unresolved adverse skin condition in the area of sensor or device placement (e.g. psoriasis, rash, Staphylococcus infection)
5. The subject has complications such as advanced autonomic neuropathy, legal blindness, or symptomatic cardiovascular disease as evidenced by a cardiovascular episode within the last six months.
6. The subject has any major concomitant disease or any physical or psychological disorder within the last five years, which might be considered life threatening or which might confound the collection or interpretation of the study data.
7. The subject has experienced two or more severe hypoglycemic events - seizures/coma requiring assistance in the past 6 months.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Comparative analysis of performance characteristics | 4 months
  Sensor clinical accuracy will be evaluated based on the following parameters: Mean ARD (absolute relative difference), median ARD, Clarke Grid Analysis. Meter BG values will be used as reference. Descriptive statistics will be used to assess non-inferiority of the Integrated sensor and infusion set sensors compare to control Enlite sensors.
Gluco-dynamic effect | 4 months
  Insulin delivery functionality will be evaluated based on BG profiles obtained during peri-prandial periods during which BG measurements will be performed at 15, 20, 30 min intervals according to the SMBG schedule. Post-prandial pharmacodynamic profiles will be analyzed to demonstrate the effect of insulin delivered using the Integrated sensor and infusion set. Specifically, rise in glucose levels followed by their fall will be used as an indication that insulin was delivered and absorbed. Post-prandial BG areas under the curve (AUC), Tmax (time to maximum rise of BG), and Cmax (maximum post-prandial BG) values will be calculated for each meal (breakfast, lunch, and dinner) consumed during both inpatient days (visits 3 and 4) and compared. Intra - and inter-subject mean values and standard deviations will be calculated. Paired and unpaired T-tests will be used to evaluate statistical significance.
Performance longevity | 4 months
  Longevity of device performance will be assessed by comparing the listed parameters obtained during visits 3 and 4.

SECONDARY OUTCOMES:
Skin condition | 4 months
  Skin condition after removal of the device will be evaluated and assessed by the clinical staff in a study survey
Physical duration | 4 months
  Investigational Center and subject's report on physical duration of the device assessed in study survey Subjects' experiences are gathered in study surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Noergaard, MDD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre Hospital, Hvidovre, Hvidovre, Denmark